CLINICAL TRIAL: NCT00706797
Title: An Open-Label, Randomized Study to Evaluate the Radiographic Efficacy and Safety of Enbrel™ (Etanercept) Added to Methotrexate in Comparison With Usual Treatment in Subjects With Moderate Rheumatoid Arthritis Disease Activity
Brief Title: Study Evaluating Efficacy / Safety of Etanercept + Methotrexate Compared to Usual Treatment in Moderate RA Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0881X1-4437
Record Dates: First submitted 2008-06-25; First posted 2008-06-30 (Estimated); Results first posted 2011-01-10 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Moderate Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Utilized Disease-Modifying Antirheumatic Drugs (DMARDs) from a list of the 6 most commonly prescribed in the participating countries (Methotrexate, sulfasalazine, hydroxychloroquine, leflunomide, cyclosporine A and gold).
  Interventions: Drug: methotrexate
- ETN + MTX (Active Comparator): Etanercept (ETN) 50 milligrams (mg) sub-cutaneous (SC) injection once weekly (pre-filled syringe) plus continuation of current dose of Methotrexate (MTX) either oral (PO), SC, or intramuscular (IM).
  Interventions: Drug: etanercept (EnbrelTM); Drug: methotrexate

INTERVENTIONS:
Drug: etanercept (EnbrelTM)
  Arms: ETN + MTX
Drug: methotrexate

SUMMARY:
To assess comparative radiographic efficacy, clinical efficacy and safety of etanercept (ETN) + methotrexate (MTX) with usual disease-modifying anti-rheumatic drug (DMARD) treatment in subjects with moderate RA who were treated with MTX monotherapy, but continue to have moderate disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Meet the 1987 ACR Revised Criteria for Rheumatoid Arthritis.
* Documented evidence, confirmed by a blinded 3rd party assessor, of at least one erosion observed by X-ray at randomization based on X-ray taken at the screening visit.
* Have received MTX as stable dose for 28 days prior to the screening visit.

Exclusion Criteria:

* Previous treatment with ETN, infliximab, adalimumab, other Tumor necrosis factor (TNF) -a inhibitors, anakinra or other biological agents.
* Receipt of any DMARD, other than MTX, within 28 days before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (40):
- Czechia (2):
  - Ostrava
  - Prague
- France (7):
  - Amiens
  - Échirolles
  - Metz
  - Montpellier
  - Paris
  - Rouen
  - Tours
- Germany (6):
  - Berlin
  - Cologne
  - Frankfurt
  - Hamburg-Eilbeck
  - Homburg
  - Mainz
- Hungary (5):
  - Budapest
  - Miskolc
  - Rijeka
  - Split
  - Zagreb
- Italy (2):
  - Jesi (Ancona)
  - Reggio Calabria
- Poland (5):
  - Bytom
  - Krakow
  - Ustroń
  - Warsaw
  - Wroclaw
- Spain (7):
  - Santander, Cantabria
  - Getafe, Madrid
  - Madrid, Madrid
  - Bilbao, Vizcaya
  - Barcelona
  - Madrid
  - Valencia
- Izmir, Turkey (Türkiye)
- United Kingdom (5):
  - Cambridge, Cambs
  - Birmingham, West Midlands
  - Aintree
  - Metropolitan Borough of Wirral
  - Newcastle

REFERENCES:
- [Derived] Mandl P, Balint PV, Brault Y, Backhaus M, D'Agostino MA, Grassi W, van der Heijde D, de Miguel E, Wakefield RJ, Logeart I, Dougados M. Clinical and ultrasound-based composite disease activity indices in rheumatoid arthritis: results from a multicenter, randomized study. Arthritis Care Res (Hoboken). 2013 Jun;65(6):879-87. doi: 10.1002/acr.21913. PMID 23213004
- [Derived] Mandl P, Balint PV, Brault Y, Backhaus M, D'Agostino MA, Grassi W, van der Heijde D, de Miguel E, Wakefield RJ, Logeart I, Dougados M. Metrologic properties of ultrasound versus clinical evaluation of synovitis in rheumatoid arthritis: results of a multicenter, randomized study. Arthritis Rheum. 2012 Apr;64(4):1272-82. doi: 10.1002/art.33491. Epub 2011 Nov 30. PMID 22131049

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 141 participants were randomized, 1 participant performed all the planned visits, and 140 participants were discontinued before completion of the study; 115 participants prematurely withdrew due to discontinuation of the study by the sponsor.
Period: Overall Study
Arm/Group | Usual Care | ETN + MTX
Started | 70 | 71
Safety Population | 63 (Safety population=all randomly assigned subjects who had at least 1 dose of study treatment.) | 71
Completed | 1 | 0
Not Completed | 69 | 71
Not completed — Lack of Efficacy | 3 | 0
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 8 | 1
Not completed — Death | 1 | 0
Not completed — Discontinuation of study by sponsor | 52 | 63
Not completed — Protocol Violation | 3 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | ETN + MTX | Total
Number analyzed (Participants) | 63 | 71 | 134
Age Continuous [Mean (Standard Deviation); unit: years] | 57.3 (12.1) | 53.8 (13.1) | 55.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 56 | 106
  Male | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Total Sharp Score (TSS) at Week 52
Description: Modified TSS is a measure of change in joint health. TSS is defined as joint space narrowing score (range 0 [no narrowing] to 168 [high narrowing]) plus (+) erosion score (range is from 0 [no erosion] to 280 [high erosion]). The modified TSS range is from 0 (no damage) to 448 (bad joint status). Increase from baseline represents disease progression and / or joint worsening; no change represents halting of disease progression; a decrease represents improvement.
Time Frame: Baseline, Week 52
Population: Modified intent-to-treat (mITT) population including all participants with an erosion at randomization confirmed by the blinded expert assessor, received at least 1 dose of subject treatment, and had data for randomization and 1 post randomization X-ray. Efficacy data not analyzed due to early termination of the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in Erosions at Week 52
Description: Erosion score (a component of the modified TSS) is a measure of change in joint health. Erosion score range is from 0 (no erosion) to 280 (high erosion). Increase from baseline represents disease progression and / or joint worsening; no change represents halting of disease progression; a decrease represents improvement.
Time Frame: Baseline, Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Joint Space Narrowing at Week 52
Description: Joint space narrowing score (a component of the modified TSS) is a measure of change in joint health. Joint space narrowing score range is 0 (no narrowing) to 168 (high narrowing). Increase from baseline represents disease progression and / or joint worsening; no change represents halting of disease progression; a decrease represents improvement.
Time Frame: Baseline, Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants Showing no Radiographic Progression (TSS Change <0.5) at Week 52
Description: Radiographic non-progression determined based on TSS change <0.5 using the dichotomous response Yes / No. The modified TSS range is from 0 (no damage) to 448 (bad joint status). Increase from baseline represents disease progression and / or joint worsening; no change represents halting of disease progression; a decrease represents improvement.
Time Frame: Baseline, Week 52, Last observation carried forward (LOCF)
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants Achieving >1.2 Improvement in Disease Activity Score Based on a 28-joint Count (DAS28)
Description: Disease activity score based on 28 painful joint counts, 28 swollen joint counts, erythrocyte sedimentation rate (ESR) in millimeters per hour (mm/hr), and general health (GH) using Visual Analog Scale (VAS); range 0 (very well) to 100 (extremely bad). DAS28 score calculated as 0.56 square root (√) (28 painful joint count) + 0.28 √ (28 swollen joint count) + 0.70 (ln ESR mm/hr) + 0.014 GH; range 0 to 10. DAS28 score >5.1=higher disease activity; <3.2=low disease activity; <2.6=clinical remission. Achievement of >1.2 improvement defined as decrease in DAS28 >1.2 (change in DAS28 < -1.2).
Time Frame: Baseline, Week 12, Week 24, and Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants Achieving Remission (DAS28 <2.60)
Description: Disease activity score based on 28 painful joint counts, 28 swollen joint counts, erythrocyte sedimentation rate (ESR) mm/hr, and general health (GH) using a visual analog scale (VAS); VAS range: 0 (very well) to 100 (extremely bad). DAS28 score calculated as 0.56 √ (28 painful joint count) + 0.28 √ (28 swollen joint count) + 0.70 (ln ESR mm/hr) + 0.014 GH; range 0 to 10. DAS28 score >5.10=higher disease activity; <3.20=low disease activity; <2.60=clinical remission.
Time Frame: Week 12, Week 24, and Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (DAS28 ≤3.20)
Description: as for outcome 6
Time Frame: Week 12, Week 24, and Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Participants Achieving a >0.6 Disease Activity Score (DAS)28 Response
Description: Disease activity score based on 28 painful joint counts, 28 swollen joint counts, erythrocyte sedimentation rate (ESR) mm/hr, and participant's assessment of general health (GH) using a visual analog scale (VAS); VAS range: 0 (very well) to 100 (extremely bad). DAS28 score calculated as 0.56 √ (28 painful joint count) + 0.28 √ (28 swollen joint count) + 0.70 (ln ESR mm/hr) + 0.014 GH; range 0 to 10. DAS28 score >5.10=higher disease activity; <3.20=low disease activity; <2.60=clinical remission. DAS28 response of >0.6 defined as decrease in DAS28 >0.6 (change in DAS28 < -0.6).
Time Frame: Week 12, Week 24, and Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percentage of Participants Achieving Moderate or Good Response on European League Against Rheumatism (EULAR) Response Criteria
Description: Response to treatment assessed by EULAR response criteria. Participants were characterized as good, moderate, or non-responders based on both Disease Activity Score (DAS) level attained and change in DAS. Good response defined as >1.2 improvement in DAS from Baseline and DAS attained during follow-up of ≤2.4. Non-responders = participants with improvement of ≤0.6 or participants with improvement of >0.6 but ≤1.2 and DAS attained during follow-up of >5.1. Remaining participants were classified as moderate. Scores of good and moderate were considered to have therapeutic response.
Time Frame: Week 12, Week 24, Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percentage of Participants With American College of Rheumatology 20% (ACR20) Response
Description: American College of Rheumatology 20% (ACR20) response: responder = ≥ 20% improvement in tender joint count; ≥ 20% improvement in swollen joint count; and ≥ 20% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and erythrocyte sedimentation rate (ESR). Subjects withdrawing early were non-responders.
Time Frame: Week 12, Week 24, Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percentage of Participants With American College of Rheumatology 50% (ACR50) Response
Description: American College of Rheumatology 50% (ACR50) response: responder = ≥ 50% improvement in tender joint count; ≥ 50% improvement in swollen joint count; and ≥ 50% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and erythrocyte sedimentation rate (ESR). Subjects withdrawing early were non-responders.
Time Frame: Week 12, Week 24, Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percentage of Participants With American College of Rheumatology 70% (ACR70) Response
Description: American College of Rheumatology 70% (ACR70) response: responder = ≥ 70% improvement in tender joint count; ≥ 70% improvement in swollen joint count; and ≥ 70% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and erythrocyte sedimentation rate (ESR) . Subjects withdrawing early were non-responders.
Time Frame: Week 12, Week 24, Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Percentage of Participants With American College of Rheumatology 90% (ACR90) Response
Description: American College of Rheumatology 90% (ACR 90) response: responder = ≥ 90% improvement in tender joint count; ≥ 90% improvement in swollen joint count; and ≥ 90% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and erythrocyte sedimentation rate (ESR). Subjects withdrawing early were non-responders.
Time Frame: Week 12, Week 24, Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline in Mean Daily Dose of Corticosteroids to Manage Flare-ups Across the 52-week Treatment Period
Description: Mean daily dose of corticosteroids to manage flare-ups (temporary increases in corticosteroid dose or use of intra-articular steroids) during treatment period. Daily dose of equivalent prednisone derived in mg/day: oral corticosteroids: 5 mg of prednisone = 5 mg of prednisolone = 25 mg of cortisone = 20 mg of hydrocortisone = 4 mg of methylprednisolone = 4 mg of triamcinolone = 2mg of paramethasone = 0.75 mg of betamethasone = 0.75 of dexamethasone = 0.3 of cortivazol.
Time Frame: Week 4, Week 12, Week 24, Week 40, Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Percentage of Participants Achieving a Minimal Clinically Important Improvement (MCII)
Description: Participants were asked how their pain had been during the last 48 hours compared to baseline. Participants that reported improvement assessed how important this improvement was to them; range: very important, moderately important, slightly important, or not at all important. Binary response options: 1=improved very important, or improved moderately important; 2=slightly important, not at all important, no change, or worse-more pain.
Time Frame: Week 12, Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Percentage of Participants Achieving a Patient Acceptable Symptom State (PASS)
Description: Percentage of participants reporting acceptable symptom state: acceptance to remain for the rest of their lives with the level of pain they had during the last 48 hours; and unacceptable symptom state: not able to remain for the rest of their lives with the level of pain they had during the last 48 hours.
Time Frame: Week 4, Week 12, Week 24, Week 40, Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Health Related Quality of Life: EuroQol-5D Health Index
Description: EQ-5D is a self-administered questionnaire to assess health-related quality of life in 5 domains (mobility, self care, usual activities, pain or discomfort, and anxiety or depression). Scores from the 5 domains are used to calculate the Health State Profile Score as a single index value; range: 0.0 (death) to 1.0 (perfect health); higher scores indicate a better health state.
Time Frame: Baseline, Week 12, Week 24, and Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Health Related Quality of Life: EuroQol-5D Health State Visual Analog Scale (VAS)
Description: EQ-5D: subject rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, Week 12, Week 24, and Week 52
Population: mITT; efficacy data not analyzed due to early termination of the study.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Usual Care | ETN + MTX
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Usual Care | ETN + MTX
Serious Adverse Events (participants affected / at risk) | 4/63 | 5/71
Other Adverse Events (participants affected / at risk) | 27/63 | 37/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=63) | ETN + MTX (N=71)
Cardiac failure (Cardiac disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Pyothorax (Infections and infestations) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=63) | ETN + MTX (N=71)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 1
Astigmatism (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 2
Myopia (Eye disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Reflux gastritis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 2
Fatigue (General disorders) | 0 | 2
Injection site erythema (General disorders) | 0 | 1
Injection site joint inflammation (General disorders) | 0 | 1
Injection site pruritus (General disorders) | 0 | 1
Injection site rash (General disorders) | 0 | 4
Injection site reaction (General disorders) | 0 | 3
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 3
Oral herpes (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 2
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 2 | 2
Viral infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Hepatitis b dna decreased (Investigations) | 0 | 1
Transaminases abnormal (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 2
Weight decreased (Investigations) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 2
Intercostal neuralgia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Urethral pain (Renal and urinary disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Thelitis (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Melanosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Thyroidectomy (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 2
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Following early termination of the study, only disposition of randomized participants, description of demographic data on safety population, and safety analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.